CLINICAL TRIAL: NCT06472999
Title: Implementation of Nephroprotective Measures in Critically Ill Patients With Moderate/Severe Acute Kidney Injury (AKI) - an Observational Study
Brief Title: Nephroprotective Measures in Critically Ill Patients With Moderate/Severe Acute Kidney Injury
Acronym: KDIGO-Bundle
Status: Recruiting | Type: Observational
Sponsor: Universität Münster (Other)
Responsible Party: Sponsor
Other Study IDs: AnIt23-10
Record Dates: First submitted 2024-06-11; First posted 2024-06-25 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; KDIGO; Nephroprotective; Bundle
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients
  Interventions: Procedure: Nephroprotective measures

INTERVENTIONS:
Procedure: Nephroprotective measures — Due to the observational design of the study, no study specific interventions are performed. The treatment of the patients is completely guided by the responsible physicians.

SUMMARY:
This study investigates to which extent recommended nephroprotective measures are implemented in critically ill patients with moderate or severe acute kidney injury.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a global problem affecting more than 10% of all hospitalized patients and up to 50% of critically ill patients, with survival related not only to the severity,1 but also to the duration of renal dysfunction.2 Recent evidence suggests that two-thirds of patients with AKI resolve their renal dysfunction within 3-7 days whereas those in whom renal dysfunctions persist have dramatically reduced survival over the following year.2 Persistence of AKI is of grave importance in that it increases an individual's risk of developing chronic kidney disease (CKD) which is a major cause of morbidity and mortality. This link between AKI and CKD has been established over the last decade3 and specific recommendations for the management of patients with AKI have been proposed in order to potentially influence this transition.4 To date, there are no specific pharmacological options for preventing or treating AKI, which is why new approaches and intensive efforts are urgently needed to reduce the occurrence of AKI. The Kidney Disease: Improving Global Outcomes (KDIGO) clinical practice guidelines recommend implementing a bundle of different supportive measures, which, in theory, should be initiated in all patients with AKI in order to prevent disease progression. However, clinical practice and recent studies have shown that the implementation of the KDIGO bundle is still not standard clinical practice despite the fact that evidence suggest clear effectiveness in the reduction of AKI rates.5-9 Poor implementation of nephroprotective measures presents a major missed opportunity to reduce AKI-related morbidity and mortality and to improve long-term outcomes. To investigate the extent to which nephroprotective measures are implemented in patients with AKI can reduce the occurrence of persistent surgical AKI, a multi-center prospective cohort study will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill patients with moderate or severe AKI (KDIGO stage 2 / 3)
2. Requirement of vasopressors or mechanical ventilation
3. Age ≥ 18 years
4. Informed consent

Exclusion Criteria:

1. Chronic kidney disease (CKD) with a glomerular filtration rate < 20ml/min
2. Chronic dialysis dependency
3. History of renal transplantation
4. Permanent ligation of the renal arteries
5. AKI immediately following nephrectomy
6. Patients requiring permanent administration of nephrotoxic drugs (e.g. immunosuppressive therapy afer liver transplantation)
7. Persons with any kind of dependency on the investigator or employed by the sponsor or investigator.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients (intensive care unit of the participating study sites)
Sampling Method: Probability Sample
Enrollment: 257 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Rate of patients in whom "Kidney Disease: Improving Global Outcomes (KDIGO)" guideline recommendations are successfully implemented for 48 hours, following the onset of moderate/ severe AKI (defined by KDIGO criteria) | 60 hours after onset of moderate/severe AKI

SECONDARY OUTCOMES:
Severity of Acute Kidney Injury | within 72 hours after diagnosis
  Severity of AKI (worst Acute Kidney Injury (AKI) stage according to Kidney Disease: Improving Global Outcomes (KDIGO) criteria, with stage 1 being the least and stage 3 being the most severe stage)
Duration of AKI (Acute Kidney Injury) | from onset of AKI until follow-up day 30
  transient AKI (< 48 hours), persistent AKI (48 hours - 7 days) or acute kidney disease (AKD) (> 7 days)

OTHER OUTCOMES:
Number of participants with recovery of baseline renal function | hospital discharge (up to 30 days)
  recovery of baseline renal function measured by estimated glomerular filtration rate (eGFR) at hospital discharge
Number of Participants with need for renal replacement therapy | within 30 days of AKI onset
  defined as whether or not any kind of renal replacement therapy became necessary at any point
Free-days of mechanical ventilation | within 30 days of AKI onset
Length of hospital stay | at hospital discharge (up to 30 days)
Length of Intensive Care Unit stay | at hospital discharge (up to 30 days)
Number of Participants with renal replacement therapy | at day 90
Mortality | at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Principal Investigator — University Münster
Locations (3):
- Universitätsklinik Innsbruck, Innsbruck, Austria
- University Hospital Münster; Department of Anesthesiology, Intensive Care Medicine and Pain Medicine, Münster, Germany
- Radboud University medical cener, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No